CLINICAL TRIAL: NCT00069342
Title: Health Beliefs and Health Behavior Practices Among Minorities With Rheumatic Diseases
Brief Title: Health Beliefs and Health Behaviors Among Minorities With Rheumatic Diseases
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 030301; 03-CC-0301
Record Dates: First submitted 2003-09-23; First posted 2003-09-24 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04-12

CONDITIONS: Rheumatoid Arthritis; Systemic Lupus Erythematosus; Arthritis
Keywords: Chronic Pain; Pain; Rheumatoid Arthritis; Depression; Function; Rheumatic Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Arthritis; Chronic Pain; Pain; Depression; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will explore the diverse health beliefs and behaviors among minority patients with rheumatic diseases. These diseases may cause joint pain, stiffness or swelling. Some can involve bones, muscles, tendons or ligaments. Some cause abnormalities of the immune system-the body's defense against disease. Some rheumatic diseases are painful or deforming and some can be life-threatening. Many rheumatic diseases occur more often and more severely in certain minority communities. This study will explore psychosocial and cultural factors related to rheumatic disease in minorities.

Patients enrolled in the NIAMS protocol Natural History or Rheumatic Disease in Minority Communities (protocol #01-AR-0227) may participate in this study. Participants will be evaluated at the NIAMS Community Health Center at the Upper Cardozo Health Center in Washington, D.C.

Participants will be interviewed about individual and community health behavior, and health beliefs about rheumatic disease and its effects on several areas of their life, including mood and physical activity. The interview will be in one of the following formats: 1) in-depth cognitive interview, 2) focus group, or 3) face-to-face interview, as follows:

In-Depth Cognitive Interview

Participants take part in a one-time interview conducted by one investigator, observed by another, and tape recorded. The interview lasts from 1 to 2 hours.

Focus Groups

Participants take part in a group interview of from 6 to 10 people during a one-time tape-recorded session that lasts from 2 to 2-1/2 hours. The group discussion is led by a moderator and a facilitator, who takes notes and makes observations.

Face-to Face Interview

Participants are interviewed twice - first upon enrollment at the NIAMS Community Health Center and again after 6 months' follow-up at the Center.

DETAILED DESCRIPTION:
Rheumatic diseases are among the most common health problems in the United States. They are a diverse group of disorders, with several shared characteristics. Marked differences in the incidence, prevalence, severity, processes of care, and outcomes in a number of rheumatic conditions exist among racial and ethnic groups as compared to white Americans. Furthermore, access to health care and treatment also differs in the minority community as compared with the majority.

The effects of the disease may be modifiable by changes in life style, diet, activities and exercise. Such changes are difficult for patients to accomplish and various strategies have been developed to facilitate success. Strategies include educational materials and programs, diet and exercise programs, patient support and empowerment programs and the like. Differences in culture and environment, lack of culturally sensitive materials and approaches, and lack of trained personnel may make these tools ineffective in the minority community. Their effectiveness in the African-American or Latino clinic population has not been assessed to date.

This is a descriptive, exploratory study designed to examine the diverse health beliefs and behaviors among the minority patients who are enrolled in the NIAMS Natural History of Rheumatic Disease in Minority Communities protocol (# 01-AR-0227). Qualitative and quantitative methodology will be used to assess the psychosocial and cultural correlates of rheumatic diseases in newly enrolled patients both at intake and after six months of being followed at the NIAMS Community Health Center, an outreach site located in the District of Columbia in the Upper Cardozo Health Center.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Phase I and II Focus Groups and Cognitive Testing of Instruments:

Previously enrolled patients with known or suspected rheumatic disease and participating in NIAMS protocol # 01-AR-0227 Natural History of Rheumatic Disease in Minority Communities Individuals identified as community leaders or members of the Community Health Partnership will also be included in the focus groups.

Phase III Baseline and Follow-up Assessments:

Newly enrolled patients (within 7 days of enrollment on protocol #01-AR-0227) with known or suspected rheumatic disease participating in NIAMS protocol # 01-AR-0227 Natural History of Rheumatic Disease in Minority Communities.

B. Age greater than or equal to 18 years.

C. Willingness and capacity to provide informed consent

EXCLUSION CRITERIA:

Patients will be excluded if any of the inclusion criteria on the parent protocol # 01-AR-0227 cannot be met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2003-09-22; Study Completion 2018-04-12

PRIMARY OUTCOMES:
Pain | Cross- Sectional

SECONDARY OUTCOMES:
functional Status -Stanford | Cross-Sectional

CONTACTS AND LOCATIONS:
Overall Officials: Gwenyth R Wallen, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wallen GR, Brooks AT. To Tell or Not to Tell: Shared Decision Making, CAM Use and Disclosure Among Underserved Patients with Rheumatic Diseases. Integr Med Insights. 2012;7:15-22. doi: 10.4137/IMI.S10333. Epub 2012 Oct 3. PMID 23071389
- [Background] Brooks AT, Andrade RE, Middleton KR, Wallen GR. Social support: a key variable for health promotion and chronic disease management in Hispanic patients with rheumatic diseases. Clin Med Insights Arthritis Musculoskelet Disord. 2014 Mar 16;7:21-6. doi: 10.4137/CMAMD.S13849. eCollection 2014. PMID 24701122